CLINICAL TRIAL: NCT02310347
Title: Influence of a Medicinal Cannabinoid Agonist on Behavioural Responses to Food Images and Food Intake: Role of Gut Peptides
Brief Title: Influence of a Medicinal Cannabinoid Agonist on Responses to Food Images and Food Intake
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S54673; 2012-003017-33 (EudraCT Number)
Record Dates: First submitted 2014-11-19; First posted 2014-12-08 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Appetite Regulation
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Marinol (Experimental): * generic name: dronabinol
  * dosage: 0.1 mg/kg
  * frequency: 2 times a single dose
  * duration: acute adminstration
  Interventions: Drug: dronabinol
- Placebo (Placebo Comparator): Empty hard gelatin capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dronabinol
  Arms: Marinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the influence of a medicinal cannabinoid agonist versus placebo on behavioural and gut peptide responses to food images and food intake.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers:

1. 20 ≤ BMI ≤ 25
2. Age 18-60
3. Right handed
4. Stable body weight for at least 3 consecutive months at start of study and no history of behavioural, therapeutic or surgical treatment aiming at or leading to weight loss/gain

For obese subjects:

1. BMI > 30
2. Age 18-60
3. Right handed
4. Stable body weight for at least 3 consecutive months at start of the study and no behavioural, therapeutic or surgical treatment aiming at or leading to weight loss/gain for at least 3 consecutive months

For FD patients:

1. FD diagnosis according to 'Rome III' criteria
2. Age 18-60
3. Right handed
4. 5% weight loss since onset of symptoms

Exclusion Criteria:

1. Medical conditions (current or history):

   * Abdominal/thoracic surgery except appendectomy
   * Gastrointestinal, endocrine (especially diabetes), or neurological diseases
   * Cardiovascular, respiratory, renal or urinary diseases
   * Hypertension
   * Food or drug allergies
   * Head trauma with loss of consciousness
2. Psychiatric disorders:

   * Eating disorders
   * Psychotic disorders
   * Major depressive disorder
   * Somatoform disorder
3. Medication use:

   * No history of cannabis use or any other drug of abuse for at least 12 months prior to the study
   * All medication except oral contraception;
4. Known allergy to dronabinol and/or sesam oil
5. Pregnancy, plans to conceive or refusal to take adequate precaution to avoid pregnancy
6. Subjects who refuse to abstain from driving during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Behavioural responses to food images and food intake | 2 years
  Scores on Visual Analogue Scales
Gut peptide responses | 2 years
  Concentrations of gut peptide levels will be determined using radioimmunoassays

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, MD, PhD, Principal Investigator — University Hospitals Leuven, campus Gasthuisberg
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Weltens N, Depoortere I, Tack J, Van Oudenhove L. Effect of acute Delta9-tetrahydrocannabinol administration on subjective and metabolic hormone responses to food stimuli and food intake in healthy humans: a randomized, placebo-controlled study. Am J Clin Nutr. 2019 Apr 1;109(4):1051-1063. doi: 10.1093/ajcn/nqz007. PMID 30949710